| Official Title: | Breast and Ovarian Catchment Pilot Grant: Clinical |
|-----------------|----------------------------------------------------|
| | Outcomes for Offering Genetic Testing in a Tiered |
| | Approach |
| NCT Number: | NCT04902144 |
| Document Type: | Study Protocol |
| Date of the | 05/15/2020 |
| Document: | |



The Human Subjects Division (HSD) strives to ensure that people with disabilities have access to all services and content. If you experience any accessibility-related issues with this form or any aspect of the application process, email hsdinfo@uw.edu for assistance.

### **INSTRUCTIONS**

- This form is only for studies that will be reviewed by the UW IRB. Before completing this form, check HSD's website to confirm that this should not be reviewed by an external (non-UW) IRB.
- <u>If you are requesting a determination</u> about whether the planned activity is human subjects research or qualifies for exempt status, you may skip all questions except those marked with a . For example 1.1 must be answered.
- Answer all questions. If a question is not applicable to the research or if you believe you have already answered a question elsewhere in the application, state "NA" (and if applicable, refer to the question where you provided the information). If you do not answer a question, the IRB does not know whether the question was overlooked or whether it is not applicable. This may result in unnecessary "back and forth" for clarification. Use non-technical language as much as possible.
- To check a box, place an "X" in the box. To fill in a text box, make sure your cursor is within the gray text box bar before typing or pasting text.
- For collaborative or multi-site research, describe only the UW activities unless you are requesting that the UW IRB provide the review and oversight for non-UW collaborators or co-investigators as well.
- You may reference other documents (such as a grant application) if they provide the requested information in non-technical language. Be sure to provide the document name, page(s), and specific sections, and upload it to **Zipline**. Also, describe any changes that may have occurred since the document was written (for example, changes that you've made during or after the grant review process). In some cases, you may need to provide additional details in the answer space as well as referencing a document.

| INDEX | | |
|---|---|---|
| 1 <u>Overview</u> | 6 Children (Minors) and Parental Permission | 10 Risk / Benefit Assessment |
| 2 Participants | 7 Assent of Children (Minors) | 11 Economic Burden to Participants |
| 3 Non-UW Research Setting | 8 Consent of Adults | 12 Resources |
| 4 Recruiting and Screening Participants | 9 Privacy and Confidentiality | 13 Other Approvals, Permissions, and<br>Regulatory Issues |
| 5 Procedures | | |

# **1 OVERVIEW**

**Study Title:** 

Breast and Ovarian Catchment Pilot Grant: Clinical Outcomes for Offering Genetic Testing in a Tiered Approach

**1.1** Home institution. Identify the institution through which the lead researcher listed on the IRB application will conduct the research. Provide any helpful explanatory information.

In general, the home institution is the institution (1) that provides the researcher's paycheck and that considers him/her to be a paid employee, or (2) at which the researcher is a matriculated student. Scholars, faculty, fellows, and students who are visiting the UW and who are the lead researcher: identify your home institution and describe the purpose and duration of your UW visit, as well as the UW department/center with which you are affiliated while at the UW.

Note that many UW clinical faculty members are paid employees of non-UW institutions.

The UW IRB provides IRB review and oversight for only those researchers who meet the criteria described in the **SOP: Use of the UW IRB**.

The lead research will conduct the research through Seattle Cancer Care Alliance.

(1.2)Consultation history. Has there been any consultation with someone at HSD about this study?

It is not necessary to obtain advance consultation. However, if advance consultation was obtained, answering this question will help ensure that the IRB is aware of and considers the advice and guidance provided in that consultation.



→ If yes, briefly describe the consultation: approximate date, with whom, and method (e.g., by email, phone call, in-person meeting).

Virtual meeting via Zoom with Jennifer McBride and Bailey Bodell from UW Reliance department on 4/24/20. Marianne Dubard-Gault (study's PI), Lauren Santos (study's research coordinator), and Martha Horik-Pyne (UW Medical Genetics research coordinator) were also present. This consultation was to discuss the involved parties of this study as well as IRB review guidance. After review, it was determined that a complete protocol application must be submitted due to the type of grant that is funding this study.

**1.3** Similar and/or related studies. Are there any related IRB applications that provide context for the proposed activities?

Examples of studies for which there is likely to be a related IRB application: Using samples or data collected by another study; recruiting subjects from a registry established by a colleague's research activity; conducting Phase 2 of a multi-part project, or conducting a continuation of another study; serving as the data coordinating center for a multi-site study that includes a UW site.

Providing this information (if relevant) may significantly improve the efficiency and consistency of the IRB's review.



→ If yes, briefly describe the other studies or applications and how they relate to the proposed activities. If the other applications were reviewed by the UW IRB, please also provide: the UW IRB number, the study title, and the lead researcher's name.

**1.4** Externally-imposed urgency or time deadlines. Are there any externally-imposed deadlines or urgency that affect the proposed activity?

HSD recognizes that everyone would like their IRB applications to be reviewed as quickly as possible. To ensure fairness, it is HSD policy to review applications in the order in which they are received. However, HSD will assign a higher priority to research with externally-imposed urgency that is beyond the control of the researcher. Researchers are encouraged to communicate as soon as possible with their HSD staff contact person when there is an urgent situation (in other words, before submitting the IRB application). Examples: a researcher plans to test an experimental vaccine that has just been developed for a newly emerging epidemic; a researcher has an unexpected opportunity to collect data from students when the end of the school year is only four weeks away.

HSD may ask for documentation of the externally-imposed urgency. A higher priority should not be requested to compensate for a researcher's failure to prepare an IRB application in a timely manner. Note that IRB review requires a certain minimum amount of time; without sufficient time, the IRB may not be able to review and approve an application by a deadline.

| X | No | |
|---|---|---|
| | Yes | → If yes, briefly describe the urgency or deadline as well as the reason for it. |

**1.5 Objectives** Using lay language, describe the purpose, specific aims, or objectives that will be met by this specific project. If hypotheses are being tested, describe them. You will be asked to describe the specific procedures in a later section.

If this application involves the use of a HUD "humanitarian" device: describe whether the use is for "on-label" clinical patient care, "off-label" clinical patient care, and/or research (collecting safety and/or effectiveness data).

This quality improvement research study aims to improve the utilization of genetic counseling and testing among providers at Olympic Medical Center (OMC) who are caring for their cancer patients in a rural and underserved area. SCCA will coach the OMC providers to offer eligible patients genetic counseling and testing in order to increase access and help the OMC site meet genetic recommendations and guidelines. Specifically, this study aims to (1) review and develop OMC's clinical operations workflow to identify cancer patients who meets criteria for genetic counseling and testing; (2) measure uptake of genetic testing; and (3) document clinical and patient reported outcomes following genetic test results.

(1.6) Study design. Provide a one-sentence description of the general study design and/or type of methodology.

Your answer will help HSD in a ssigning applications to reviewers and in managing workload. Examples: a longitudinal observational study; a double-blind, placebo-controlled randomized study; ethnographic interviews; web scraping from a convenience sample of blogs; medical record review; coordinating center for a multi-site study.

This is a quality improvement research study in which SCCA will provide coaching to OMC providers to offer genetic counseling and testing in order to address current gaps in caring for their high-risk patients.

(1.7) Intent. Check all the descriptors that apply to your activity. You must place an "X" in at least one box.

This question is essential for ensuring that your application is correctly reviewed. Please read each option carefully.



| 3. Improve the quality of service provided by a specific institution, organization, or program. |
|---|
| <ul> <li>4. Designed to expand the knowledge base of a scientific discipline or other scholarly field of study, and produce results that:</li> <li>Are expected to be applicable to a larger population beyond the site of data collection or the specific subjects studied, or</li> <li>Are intended to be used to develop, test, or support theories, principles, and statements of relationships, or to inform policy beyond the study.</li> </ul> |
| 5. Focus directly on the specific individuals about whom the information or biospecimens are collected through oral history, journalism, biography, or historical scholarship activities, to provide an accurate and evidence-based portrayal of the individuals. |
| 6. A quality improvement or program improvement activity conducted to improve the implementation (delivery or quality) of an accepted practice, or to collect data about the implementation of the practice for clinical, practical, or administrative purposes. This does not include the evaluation of the efficacy of different accepted practices, or a comparison of their efficacy. |
| 7. Public health surveillance activities conducted, requested, or authorized by a public health authority for the sole purpose of identifying or investigating potential public health signals or timely awareness and priority setting during a situation that threatens public health. |
| 8. Preliminary, exploratory, or research development activities (such as pilot and feasibility studies, or reliability/validation testing of a questionnaire) |
| 9. Expanded access use of a drug or device not yet approved for this purpose |
| 10. Use of a Humanitarian Use Device |
| 11. Other. Explain: |

- **1.8 Background, experience, and preliminary work**. Answer this question <u>only</u> if the proposed activity has one or more of the following characteristics. The purpose of this question is to provide the IRB with information that is relevant to its risk/benefit analysis.
  - Involves more than minimal risk (physical or non-physical)
  - Is a clinical trial, or
  - Involves having the subjects use a drug, biological, botanical, nutritional supplement, or medical device.

"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests.

**a.** <u>Background</u>. Provide the rationale and the scientific or scholarly background for the proposed activity, based on existing literature (or clinical knowledge). Describe the gaps in current knowledge that the project is intended to address.

This should be a plain language description. Do not provide scholarly citations. Limit your answer to less than one page, or refer to an attached document with background information that is no more than three pages long.

N/A

**b.** Experience and preliminary work. Briefly describe experience or preliminary work or data (if any) that you, your team, or your collaborators/co-investigators have that supports the feasibility and/or safety of this study.

It is not necessary to summarize all discussion that has led to the development of the study protocol. The IRB is interested only in short summaries about experiences or preliminary work that suggest the study is feasible and that risks are reasonable relative to the benefits. Examples: Your team has already conducted a Phase 1 study of an experimental drug which supports the Phase 2 study being proposed in this application; your team has already done a small pilot study showing that the reading skills intervention described in this application is feasible in an after-school program with classroom aides; your team has experience with the type of surgery that is required to implant the study device; the study coordinator is experienced in working with subjects who have significant cognitive impairment.

N/A

**1.9 Supplements**. Check all boxes that apply, to identify relevant Supplements that should be completed and uploaded to *Zipline*.

This section is here instead of at the end of the form to reduce the risk of duplicating information in this IRB Protocol form that you will need to provide in these Supplements.

| Check all<br>That Apply | Type of Research | Supplement Name |
|---|---|---|
| | <b>Department of Defense</b> The research involves Department of Defense funding, facilities, data, or personnel. | ZIPLINE SUPPLEMENT: Department of Defense |
| | Department of Energy The research involves Department of Energy funding, facilities, data, or personnel. | ZIPLINE SUPPLEMENT: Department of Energy |
| | Drug, biologic, botanical, supplement Procedures involve the use of <u>any</u> drug, biologic, botanical or supplement, even if the item is not the focus of the proposed research | ZIPLINE SUPPLEMENT: Drugs |
| | Emergency exception to informed consent Research that requires this special consent waiver for research involving more than minimal risk | ZIPLINE SUPPLEMENT: Exception from Informed Consent for Emergency Research (EFIC) |
| | Genomic data sharing | ZIPLINE SUPPLEMENT: Genomic Data Sharing |

| | | 1 |
|---|---|---|
| | Genomic data are being collected and will be deposited in an external database (such as the NIH dbGaP database) for sharing with other | |
| | researchers, and the UW is being asked to provide the required | |
| | certification or to ensure that the consent forms can be certified | |
| | Medical device | |
| | Procedures involve the use of <u>any</u> medical device, even if the device is | ZIPLINE SUPPLEMENT: |
| | not the focus of the proposed research, except when the device is FDA- | Devices |
| | approved and is being used through a clinical facility in the manner for | <u>Devices</u> |
| | which it is approved | |
| | Multi-site or collaborative study | CLIDDI ENAENT, Multi cito |
| | The UW IRB is being asked to review on behalf of one or more non-UW | SUPPLEMENT: Multi-site<br>or Collaborative Research |
| | institutions in a multi-site or collaborative study. | or conaborative research |
| | Non-UW Individual Investigators | 1 1 |
| | The UW IRB is being asked to review on behalf of one or more non-UW | SUPPLEMENT: Non-UW |
| | individuals who are not affiliated with another organization for the | Individual Investigators |
| | purpose of the research. | |
| Х | None of the above | |

# **2 PARTICIPANTS**

**(2.1)**Participants. Describe the general characteristics of the subject populations or groups, including age range, gender, health status, and any other relevant characteristics.

The subject groups for this study will consist of OMC medical oncology providers and OMC patients between 19-90 years old with a diagnosis of cancer.

- (2.2) Inclusion and exclusion criteria.
  - **a. Inclusion criteria.** Describe the specific criteria that will be used to decide who will be included in the research from among interested or potential subjects. Define any technical terms in lay language.

Participants will include medical oncology providers at OMC who see patients with an active diagnosis of breast, ovarian, prostate, colon, or pancreatic cancer. The OMC providers will be consenting to release their patients' medical records to SCCA so that SCCA subject matter experts (cancer geneticist and/or genetic counselor) can identify patients with an underlying hereditary cancer syndrome to be offered genetic counseling and testing.

**b. Exclusion criteria.** Describe the specific criteria that will be used to decide who will be excluded from the research from subjects who meet the inclusion criteria listed above. Define any technical terms in lay language.

This study will exclude OMC providers who do not see patients with an active diagnosis of cancer. This study will exclude patients who are minors, patients without an active diagnosis of cancer, and patients with precancerous lesions such as ductal carcinoma in situ (the presence of abnormal cells inside a milk duct in the breast) or colon polyps (a small clump of cells that form on the lining of the colon or rectum).

2.3) Prisoners. IRB approval is required in order to include prisoners in research, even when prisoners are not an intended target population. a. Will the proposed research recruit or obtain data from individuals that are known to be prisoners? For records reviews: if the records do not indicate prisoner status and prisoners are not a target population, select "No". See the WORKSHEET: Prisoners for the definition of "prisoner".  $\rightarrow$  If no, skip the rest of part a. and continue to 2.3.b **Yes**  $\rightarrow$  If yes, answer the following questions (i – iv). i. Describe the type of prisoners, and which prisons/jails: ii. One concern about prisoner research is whether the effect of participation on prisoners' general living conditions, medical care, quality of food, amenities, and/or opportunity for earnings in prison will be so great that it will make it difficult for prisoners to adequately consider the research risks. How will the chances of this be reduced? iii. Describe what will be done to make sure that (a) recruitment and subject selection procedures will be fair to all eligible prisoners and (b) prison authorities or other prisoners will not be able to arbitrarily prevent or require particular prisoners from participating. iv. If the research will involve prisoners in federal facilities or in state/local facilities outside of Washington State: check the box below to provide assurance that study team members will (a) not encourage or facilitate the use of a prisoner's participation in the research to influence parole decisions, and (b) clearly inform each prisoner in advance (for example, in a consent form) that participation in the research will have no effect on his or her parole. Confirmed **b.** Is the research likely to have subjects who become prisoners while participating in the study? For example, a longitudinal study of youth with drug problems is likely to have subjects who will be prisoners at some point during the study. No → If yes, if a subject becomes a prisoner while participating in the study, will any study Yes procedures and/or data collection related to the subject be continued while the subject is a prisoner? No

→ If yes, describe the procedures and/or data collection that will continue with

prisoner subjects

Yes

Version 2.2

**2.4)Protected populations**. IRB approval is required for the use of the subject populations listed here. Check the boxes for any of these populations that will be purposefully included. (In other words, being a part of the population is an inclusion criterion for the study.)

The WORKSHEETS describe the criteria for approval but do not need to be completed and should not be submitted.

| Population | Worksheet |
|---------------------------------|---------------------------|
| Fetuses in utero | WORKSHEET: Pregnant Women |
| Neonates of uncertain viability | WORKSHEET: Neonates |
| Non-viable neonates | WORKSHEET: Neonates |
| Pregnant women | WORKSHEET: Pregnant Women |

a. If you check any of the boxes above, use this space to provide any information that may be relevant for the IRB to consider.

None of the populations listed above will be purposefully included in this study.

**2.5)Native Americans or non-U.S. indigenous populations.** Will Native American or non-U.S. indigenous populations be actively recruited through a tribe, tribe-focused organization, or similar community-based organization?

Indigenous people are defined in international or national legislation as having a set of specific rights based on their historical ties to a particular territory and their cultural or historical distinctiveness from other populations that are often politically dominant.

Examples: a reservation school or health clinic; recruiting during a tribal community gathering

Yes

→ If yes, name the tribe, tribal-focused organization, or similar community-based organization. The UW IRB expects that tribal/indigenous approval will be obtained before beginning the research. This may or may not involve approval from a tribal IRB. The study team and any collaborators/investigators are also responsible for identifying any tribal laws that may affect the research.

**2.6) Third party subjects.** Will the research collect private identifiable information about other individuals from the study subjects? Common examples include: collecting medical history information or contact information about family members, friends, co-workers.

"Identifiable" means any direct or indirect identifier that, alone or in combination, would allow you or another member of the research team to readily identify the person. For example, suppose that the research is about immigration history. If subjects are asked questions about their grandparents but are not asked for names or other information that would allow easy identification of the grandparents, then private identifiable information is not being collected about the grandparents and the grandparents are not subjects.

No

**Document Date & Version** 11/15/2019 Version 2.2

#2003

| Yes → If yes, these individuals are considered huma will be collected about them. | n subjects in the study. Describe them and what data |
|---|---|
| <b>2.7 Number of subjects.</b> Is it possible to predict or describe the m needed to complete the study, for each subject group? | naximum number of subjects (or subject units) |
| Subject units mean units within a group. For most research studies, interest in some research is not the individual. Examples: Dyads such as caregiver-and-Alzheimer's patient, or parent Families Other units, such as student-parent-teacher Subject group means categories of subjects that are meaningful for group — for example, all UW students taking Introductory Psycholog | t and child the specific study. Some research has only one subject |
| <ul> <li>include:</li> <li>By intervention – for example, an intervention group and a</li> <li>By subject population or setting – for example, urban versu</li> <li>By age – for example, children who are 6, 10, or 14 years of</li> </ul> | ıs rural families |
| The IRB reviews the number of subjects in the context of risks and be that the research involves no more than minimal risk: there are no renrolled. If the research involves more than minimal risk: The number described in this application. If it is necessary later to increase the number (over-enrollment) will be considered non-composite the provided the rationale in the box below. A the scope/size of the research. You do not need | restrictions on the total number of subjects that may be er of enrolled subjects must be limited to the number number of subjects, submit a Modification. Exceeding the appliance. Also, provide any other available information about |
| Example: It may not be possible to predict the number advertised through Craigslist, but you can state that who respond is the number who will be in the study | t the survey will be posted for two weeks and the number |
| | low to provide the estimate of the maximum desired uch as families) who will complete the research. |
| Group name/description | Maximum desired number of individuals (or other subject unit, such as families) who will complete the research Provide numbers for the site(s) reviewed by the UW IRB and for the study-wide total number; example: 20/100 |
| OMCillilililii | |
| OMC providers who see patients with an active diagnosis of breast, ovarian, prostate, colon, or pancreatic cancer | 6 (4 MDs, 1 PA-C, and 1 ARNP) |
| Phase 1: Patients in the observational group in which SCCA collects data on OMC patients who follow their current processes (without intervention) | 60/120 |

Document Date & Version \_\_\_\_\_\_ Dubard-Gault

60/120

Phase 2: Patients in the monitoring group in which SCCA collect data on OMC patients who follow the tiered

intervention (OMC providers receive coaching from

SCCA subject matter experts)

# **3 NON-UW RESEARCH SETTING**

Complete this section only if UW investigators and people named in the <u>SUPPLEMENT:</u>
<u>Non-UW Individual Investigators</u> will conduct research procedures outside of UW and Harborview

**3.1**) Reason for locations. Describe the reason(s) for choosing the locations.

This is especially important when the research will occur in locations or with populations that may be vulnerable to exploitation. One of the three ethical principles the IRB must consider is justice: ensuring that reasonable, non-exploitative, and well-considered procedures are administered fairly, with a fair distribution of costs and potential benefits.

OMC is the ideal site for this research study because of its rural and underserved location, which can pose many obstacles to their patients in accessing genetic evaluations for the treatment of their cancers and for their family members. OMC is an affiliate site of SCCA and this partnership, in which SCCA will provide coaching to OMC providers, will facilitate a more open line of communication between the sites. OMC providers will have the resources to increase access to genetic counseling and testing to its patients as well as refer their patients with more complicated cases to SCCA for genetic consultation services

**3.2** Local context. Culturally appropriate procedures and an understanding of local context are an important part of protecting subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect the research, how it is conducted, or how consent is obtained or documented.

Examples: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male researcher; instead, the researcher may need to ask a male family member for permission before the woman can be approached. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual members of a group. In some distinct cultural groups, signing forms may not be the norm.

This federal site maintains an international list of human research standards and requirements: <a href="http://www.hhs.gov/ohrp/international/index.html">http://www.hhs.gov/ohrp/international/index.html</a>

N/A

- **3.3** Location-specific laws. Describe any local laws that may affect the research (especially the research design and consent procedures). The most common examples are laws about:
  - **Specimens** for example, some countries will not allow biospecimens to be taken out of the country.
  - **Age of consent** laws about when an individual is considered old enough to be able to provide consent vary across states, and across countries.
  - Legally authorized representative laws about who can serve as a legally authorized representative (and who has priority when more than one person is available) vary across states and countries.
  - **Use of healthcare records** many states (including Washington State) have laws that are similar to the federal HIPAA law but that have additional requirements.

N/A. OMC is located in Sequim, Washington. The laws in this region are the same as the laws that apply to SCCA.

Document Date & Version 11/15/2019 Version 2.2 #2003 **Dubard-Gault** 

that affect the research.

Example: A school district may require researchers to obtain permission from the head district office as well as school principals before approaching teachers or students; a factory in China may allow researchers to interview factory workers but not allow the workers to be paid for their participation.

N/A

3.5 If the PI is a student: Does the research involve traveling outside of the US?

No

Yes 

If yes, confirm by checking the box that (1) you will register with the UW Office of Global Affairs before traveling; (2) you will notify your advisor when the registration is complete; and (3) you will request a UW Travel Waiver if the research involves travel to the list of countries requiring a UW

3.4)Location-specific administrative or ethical requirements. Describe local administrative or ethical requirements

# 4 RECRUITING and SCREENING PARTICIPANTS

Confirmed

Travel Waiver.

**4.1** Recruiting and Screening. Describe how subjects will be identified, recruited, and screened. Include information about: how, when, where, and in what setting. Identify who (by position or role, not name) will approach and recruit subjects, and who will screen them for eligibility.

Before the study begins, the SCCA study team will identify OMC providers who meet eligibility criteria through the OMC website's oncology providers page. A virtual meeting (via Zoom) will be set up by the study's research coordinator to include the SCCA study team and OMC's medical director and all the potential OMC provider subjects. During this meeting, the PI and research coordinator will explain the study's target patient population, methods, procedures, and goals. OMC providers will be given time to introduce themselves and describe their patient population to ensure that they are eligible to participate.

#### 4.2 Recruitment materials.

a. What materials (if any) will be used to recruit and screen subjects?

Examples: talking points for phone or in-person conversations; video or audio presentations; websites; social media messages; written materials such as letters, flyers for posting, brochures, or printed advertisements; questionnaires filled out by potential subjects.

The SCCA study team will recruit all eligible OMC providers via a virtual meeting (through Zoom), where the study will be described and discussed in detail. As part of recruitment, all potential OMC provider participants will be provided copies of the study's research methods and procedures. After this meeting, the study's research coordinator will then email a consent information sheet (attached in Zipline). The OMC providers who choose to participant will send an emailed consent to the study's research coordinator.

There is no recruitment process for OMC patients because the study team will have no contact with the patients at any point of the study. OMC patients will be screened by reviewing their clinical diagnosis and stage, pathology report features, and treatment options (after consent is given from their OMC provider to release their medical records).

**b.** Upload descriptions of each type of material (or the materials themselves) to **Zipline**. If letters or emails will be sent to any subjects, these should include a statement about how the subject's name and contact information were obtained. No sensitive information about the person (such as a diagnosis of a medical condition) should be included in the letter.

HSD encourages researchers to consider uploading descriptions of most recruitment and screening materials instead of the materials themselves. The goal is to provide the researchers with the flexibility to change some information on the materials without submitting a Modification for IRB approval of the changes. Examples:

- Provide a list of talking points that will be used for phone or in-person conversations instead of a script.
- For the description of a flyer, include the information that it will provide the study phone number and the name of a study contact person (without providing the actual phone number or name). This means that a Modification would not be necessary if/when the study phone number or contact person changes. Also, instead of listing the inclusion/exclusion criteria, the description below might state that the flyer will list one or a few of the major inclusion/exclusion criteria.
- For the description of a video or a website, include a description of the possible visual elements and a list of the content (e.g., study phone number; study contact person; top three inclusion/exclusion criteria; payment of \$50; study name; UW researcher).
- **4.3 Relationship with participant population**. Do any members of the study team have an existing relationship with the study population(s)?

Examples: a study team member may have a dual role with the study population (for example, being their clinical care provider, teacher, laboratory directory or tribal leader in addition to recruiting them for his/her research).



No Yes

→ If yes, describe the nature of the relationship.

**4.4 Payment to participants**. Describe any payment that will be provided, including:

- The total amount/value
- Whether payment will be "pro-rated" so that participants who are unable to complete the research may still receive some part of the payment

The IRB expects the consent process or study information provided to the subjects to include information about the number and amount of payments, and especially the time when subjects can expect to receive payment. One of the most frequent complaints received by HSD is from subjects who expected to receive cash or a check on the day that they completed a study and who were angry or disappointed when payment took 6-8 weeks to reach them.

Do not include a description of any expenses that will be reimbursed.

No payment will be provided to participants.

**4.5** Non-monetary compensation. Describe any non-monetary compensation that will be provided. Example: extra credit for students; a toy for a child. If class credit will be offered to students, there must be an alternate way for the students to earn the extra credit without participating in the research.

No non-monetary compensation will be provided to participants.

| | Yes → If yes, describe the data an the study data. | d/or specimens (including PHI) and whether it will be retained as part of |
|---|---|---|
| 1.7 | | ll consent be obtained for any of the recruiting and screening asks about consent for the main study procedures). |
| | | for their own participation; parental permission; assent from children; consent dult individuals who are unable to provide consent. |
| | <ul> <li>from the registry participants to relect</li> <li>For a study in which possible subjects</li> <li>For a study in which individuals response</li> </ul> | |
| | ' | ent. Will a written or verifiable electronic signature from the subject on a odocument consent for the recruiting and screening procedures? |
| | I INO | cribe the information that will be provided during the consent process which procedures. |
| | Yes → If yes, up | load the consent form to <b>Zipline</b> . |
| 5 1 | 5 PROCEDURES | |
| 5.1 | , | ovide a complete description of the study procedures, including the if any), drug dosing information (if any), use of records, time required, bad a study flow sheet or table to <i>Zipline</i> . |
| | Risks of Harm from Standard Care and the dr | important to accurately identify the research procedures. See UW IRB <u>POLICY:</u> aft guidance from the federal Office of Human Research Protections, <u>"Guidance"</u> in Research Evaluating Standards of Care"; October 20, 2014. |

(4.6) Will data or specimens be accessed or obtained for recruiting and screening procedures prior to enrollment?

 $\rightarrow$  If no, skip the rest of this section; go to <u>question 5.1</u>.

Examples: names and contact information; the information gathered from records that were screened; results of screening questionnaires or screening blood tests; Protected Health Information (PHI) from screening medical records to identify possible

subjects.

Dubard-Gault

This quality improvement research study is designed in two phases, each phase is done over a 3-month period for a total study duration of 6 months. The SCCA study team will be enrolling eligible OMC providers who will handle all patient interaction and communication.

Phase 1: The first phase does not involve intervention; OMC will be following their existing processes. OMC will gather identified data on the patient's clinic diagnosis and stage, pathology report features, and treatment options for patients with the above diagnose and offer patients the option to fill out a standardized Family History Questionnaire (FHQ) on the day of their initial visit if they decide to do so. The FHQ will be offered as part of clinical care up to the discretion of the OMC providers. OMC will also gather de-identified data on the number of patients seen with a diagnosis of breast, ovarian, prostate, colon, and pancreatic cancer. The above data will then be sent to the study's research coordinator at SCCA (through secure email) which will be stored in a secured J-Drive folder within the SCCA network. The research coordinator will randomly assign all identified patient data to a unique participant ID before distributing to SCCA subject matter experts (cancer geneticist and/or genetic counselor) for review. From OMC's collected data, SCCA subject matter experts will measure how many patients met NCCN criteria for testing how many patients were referred to genetic counseling and how many either had a test online or were seen at UWMC and the SCCA for a genetic evaluation.

Phase 2: The second phase involves a tiered intervention in which SCCA subject matter experts will coach the OMC providers to provide guidance on providing genetic counseling and testing to their patients. Involvement in this study does not dictate how the OMC providers carry out clinical care, so it is up to the OMC providers to decide whether or not to implement the coaching in their practice. First, patients and their families fill out the standardized FHQ before their initial appointment, which will be sent via email by the team at OMC. OMC will gather the same patient information described in Phase 1 which will then be sent directly to the study's research coordinator at SCCA, where the research coordinator will follow the same data storage, participant ID assignment, and distribution processes as in Phase 1. SCCA subject matter experts would then review this information with the OMC providers at bi-monthly virtual conferences before patients come for their initial visit at OMC. For patients who meet NCCN criteria, the oncology team at OMC would include in their initial visit workflow to discuss importance of cancer risk assessment and offer genetic testing. For the patients with a more complicated history, the OMC team would offer a referral to the SCCA for a complete cancer risk assessment evaluation.

At the end of phase 2, SCCA subject matter experts will measure how many patients met NCCN criteria for testing how many patients were referred to genetic counseling and how many either had a test online or were seen at UWMC and the SCCA for a genetic evaluation. This data will then be compared with phase 1 data to measure the effectiveness of SCCA's coaching for OMC's providers as well as quality improvement of their processes.

(5.2 Recordings. Does the research involve creating audio or video recordings?

| X No | → If no, go to question 5.3. |
|---|---|
| Yes | → If yes, describe what will be recorded (if not already described in 5.1) and answer question <b>a</b> . |
| | a. Before recording, will consent for being recorded be obtained from subjects and any other<br>individuals who may be recorded? |
| | No → If no, email <a href="mailto:hsdinfo@uw.edu">hsdinfo@uw.edu</a> before submitting this application in Zipline. In the email, include a brief description of the research and a note that individuals will be recorded without their advance consent. |
| | Yes |
| 5.3 MRI scans. | Will any subjects have a Magnetic Resonance Imaging (MRI) scan as part of the study procedures? |

This means scans that are performed solely for research purposes or clinical scans that are modified for research purposes (for example, using a gadolinium-based contrast agent when it is not required for clinical reasons).

**X** No  $\rightarrow$  If no, go to question 5.4.

| _ | |
|-----|---------------------------------------------|
| Yes | → If yes, answer questions <b>a</b> through |
| | a. Describe the MRI scan(s). Specifically |

- What is the purpose of the scan(s)? Examples: obtain research data; safety assessment associated with a research procedure.
- Which subjects will receive an MRI scan?
- Describe the minimum and maximum number of scans per subject, and over what time period the scans will occur. For example: all subjects will undergo two MRI scans, six months apart.

| b. Use of gadolinium. | Will any of the MRI scans involve the use of a gadolinium-based contrast agent |
|---|---|
| (GBCA?) | |

| N |
|----|
| Ye |

→ If yes, which agents will be used? Check all that apply.

| Brand Name | Generic Name | Chemical Structure |
|----------------------|--------------------------|--------------------|
| Dotarem | Gadoterate meglumine | Macrocylic |
| Eovist / Primovist | Gadoxetate disodium | Linear |
| Gadavist | Gadobutro | Macrocyclic |
| Magnevist | Gadpentetate dimeglumine | Linear |
| MultiHance | Gadobenate dimeglumine | Linear |
| Omniscan | Gadodiamide | Linear |
| OptiMARK | Gadoversetamide | Linear |
| ProHance | Gadoteridol | Macrocyclic |
| Other, provide name: | | |

1.) The FDA has concluded that gadolinium is retained in the body and brain for a significantly longer time than previously recognized, especially for linear GBCAs. The health-related risks of this longer retention are not yet clearly established. However, the UW IRB expects researchers to provide a compelling justification for using a linear GBCA instead of a macrocyclic GBCA, to manage the risks associated with GBCAs.

Describe why it is important to use a GBCA with the MRI scan(s). Describe the dose that will be used and (if it is more than the standard clinical dose recommended by the manufacturer) why it is necessary to use a higher dose. If a linear GBCA will be used, explain why a macrocyclic GBCA cannot be used.

2.) Information for subjects. Confirm by checking this box that subjects will be provided with the FDA-approved Patient Medication Guide for the GBCA being used in the research or that the same information will be inserted into the consent form.

| - |
|-------------|
| C |
| l Confirmed |

c. MRI facility. At which facility(ies) will the MRI scans occur? Check all that apply.

| UWMC Radiology/Imaging Services (the UWMC clinical facility) |
|--------------------------------------------------------------------------|
| DISC Diagnostic Imaging Sciences Center (UWMC research facility) |
| BMIC Biomolecular Imaging Center (South Lake Union research facility) |
| Harborview Radiology/Imaging Services (the Harborview clinical facility) |
| SCCA Imaging Services |
| Northwest Diagnostic Imaging |
| Other: identify in the text box below: |

**Personnel.** For MRI scans that will be conducted at the DISC or BMIC research facilities: The role, qualifications, and training of individuals who will operate the scanner, administer the GBCA (if applicable), and/or insert and remove the IV catheter should be described in question **12.3**.

(5.4) Data variables. Describe the specific data that will be obtained (including a description of the most sensitive items). Alternatively, a list of the data variables may be uploaded to *Zipline*.

OMC clinic outcomes data: report including the number of patients seen at OMC with a diagnosis of breast, ovarian, prostate, colon, and pancreatic cancer

OMC patients' Family History Questionnaire responses

OMC patients' identified data on clinical diagnosis and stage, pathology report features, and treatment options for patients with a diagnosis of breast, ovarian, prostate, colon, and pancreatic cancer

**5.5 Data sources.** For all types of data that will be accessed or collected for this research: Identify whether the data are being obtained from the subjects (or subjects' specimens) or whether they are being obtained from some other source (and identify the source).

If you have already provided this information in Question 5.1, you do not need to repeat the information here.

OMC clinic outcomes data: pulled from patients' clinical charts e.g. "referred for genetic counseling". Collected by OMC

Family History Questionnaire responses: filled out directly by patients then collected by OMC OMC patients' identified data/relevant medical records: pulled from Epic. Collected by OMC

**5.6** Identifiability of data and specimens. Answer these questions carefully and completely. This will allow HSD to accurately determine the type of review that is required and the relevant compliance requirements. Review the following definitions before answering the questions:

Access means to view or perceive data, but not to possess or record it. See, in contrast, the definition of "obtain".

Identifiable means that the identity of an individual is or may be readily (1) ascertained by the researcher or any other member of the study team from specific data variables or from a combination of data variables, or (2) associated with the information.

Direct identifiers are direct links between a subject and data/specimens. Examples include (but are not limited to): name, date of birth, medical record number, email or IP address, pathology or surgery accession number, student number, or a collection of data that is (when taken together) identifiable.

**Indirect identifiers** are information that links between direct identifiers and data/specimens. Examples: a subject code or pseudonym.

**Key** refers to a single place where direct identifiers and indirect identifiers are linked together so that, for example, coded data can be identified as relating to a specific person. Example: a master list that contains the data code and the identifiers linked to the codes.

**Obtain** means to possess or record in any fashion (writing, electronic document, video, email, voice recording, etc.) for research purposes and to retain for any length of time. This is different from **accessing**, which means to view or perceive data.

| a. Will you or any members of your team have access to any direct or indirect identifiers? | |
|---|---|
| X Yes | If yes, describe which identifiers and for which data/specimens. |
| | OMC will have access to all of their patients' identifiers as part of their standard processes of care. The SCCA study team will not have direct access to any direct or indirect identifiers unless sent to them by OMC. |
| No | → If no, select the reason(s) why you (and all members of your team) will not have access to direct or indirect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before access. |
| There is an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to study team members under any circumstances. | |
| This agreement should be available upon request from the IRB. Examples: a Data Use Agree Repository Gatekeeping form, or documented email. | |
| There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link includes situations involving an Honest Broker. | |
| | There are other legal requirements prohibiting the release of the identifiers or key. Describe them below. |

Version 2.2

| <b>b.</b> Will you or any study team members <u>obtain</u> any direct or indirect identifiers? | |
|---|---|
| X Yes → If yes, describe which identifiers and for which data/specimens. | |
| | The study's research coordinator will obtain identifiers through OMC as included in the patients' medical records. This will include medical record number, first and last name, and date of birth. |
| No → If no, select the reason(s) why you (and all members of your team) will not obtain direct indirect identifiers. | |
| | There will be no identifiers. |
| _ | Identifiers or the key have been (or will have been) destroyed before access. |
| [ | There will be an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) under any circumstances. |
| _ | This agreement should be available upon request from the IRB. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). The includes situations involving an Honest Broker. | |
| There are other legal requirements prohibiting the release of the identifiers or key. Describe them below. | |
| • | will be obtained, indicate how the identifiers will be stored (and for which data). NOTE: Do<br>data security plan here – that information is requested in section 9.6. |
| [ | Identifiers will be stored with the data. Describe the data to which this applies: |
| _ | |
| Ε | Identifiers and study data will be stored separately but a link will be maintained between the identifiers and the study data (for example, through the use of a code). Describe the data to which this applies: |
| _ | This will apply to FHQ results as well as data on patients' clinical diagnosis and stage, pathology report features, and treatment options. The study's research coordinator will use a tracking sheet to document patient identification and their assigned participant ID, which will be stored in a private SCCA network J-drive folder. |
| | Identifiers and study data will be stored separately, with no link between the identifiers and the study data. Describe the data to which this applies: |

**d. Research collaboration**. Will individuals who provide coded information or specimens for the research also collaborate on other activities for this research? If yes, identify the activities and provide the name of the collaborator's institution/organization.

Examples include but are not limited to: (1) study, interpretation, or analysis of the data that results from the coded information or specimens; and (2) authorship on presentations or manuscripts related to this work.

Yes: The study's research coordinator will be involved in coordinating and organizing the bi-monthly conference meetings with the OMC provider subjects and SCCA study team. They will also be involved in the interpretation and analysis of the data that results from the coded information.

(5.7) Protected Health Information (PHI). Will participants' identifiable PHI be accessed, obtained, used, or disclosed for any reason (for example, to identify or screen potential subjects, to obtain study data or specimens, for study follow-up) that does not involve the creation or obtaining of a Limited Data Set?

PHI is individually identifiable healthcare record information or clinical specimens from an organization considered a "covered entity" by federal HIPAA regulations, in any form or media, whether electronic, paper, or oral. You must answer yes to this question if the research involves identifiable health care records (e.g., medical, dental, pharmacy, nursing, billing, etc.), identifiable healthcare information from a clinical department repository, or observations or recordings of clinical interactions.

X Yes

→ If no, skip the rest of this question; go to question 5.8

→ If yes, answer all of the questions below.

**a.** Describe the PHI and the reason for using it. Be specific. For example, will any "free text" fields (such as physician notes) be accessed, obtained, or used?

PHI will include patient's free text medical records regarding their clinical diagnosis and stage, pathology report features, and treatment options. It will also include their responses to the FHQ. This identified information will be accessed and obtained by OMC and the study's research coordinator at SCCA. The research coordinator will need access to the identified data in order to ensure seamless communication between OMC oncologists and the SCCA subject matter experts during meetings to identify and provide coaching on eligible patients for genetic counseling and testing.

**b.** Is any of the PHI located in Washington State?

No X Yes

**c.** Describe the pathway of how the PHI will be accessed or obtained, starting with the source/location and then describing the system/path/mechanism by which it will be identified, accessed, and copied for the research. Be specific. For example: directly view records; search through a department's clinical database; submit a request to Leaf.

OMC will directly access PHI through their medical records system. These will be compiled into patient packets as a single PDF for each, which will then be sent via secure email to the study's research coordinator at SCCA. The research coordinator will then securely store this information within a private SCCA network J-drive folder.

**d.** For which PHI will subjects provide HIPAA authorization before the PHI is accessed, obtained and/or used?

N/A. Subjects will not provide HIPAA authorization for any PHI

<u>Confirm by checking the box</u> that the UW Medicine <u>HIPAA Authorization</u> form maintained on the HSD website will be used to access, obtain, use, or disclose any UW Medicine PHI.

Confirmed

Document Date & Version 11/15/2019 Version 2.2 #2003

ZIPLINE APPLICATION: IRB Protocol

e. For which PHI will HIPAA authorization NOT be obtained from the subjects?

HIPAA authorization will not be obtained for any PHI from the OMC patient subjects. OMC has an established connection with SCCA as an SCCA affiliate site and already transfers patients' medical records to SCCA oncologists for review/second opinion. Transfer of PHI within the study will follow those same established guidelines.

Provide the following assurances by checking the boxes.

The minimum necessary amount of PHI to accomplish the purposes described in this application will be accessed, obtained and/or used.

The PHI will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research study, or for other research for which the use or disclosure of PHI would be permitted.

The HIPAA "accounting for disclosures" requirement will be fulfilled, if applicable. See <a href="UW">UW</a> <a href="Medicine Compliance Policy #104">Medicine Compliance Policy #104</a>.

There will be reasonable safeguards to protect against identifying, directly or indirectly, any patient in any report of the research.

**5.8** Genomic data sharing. Will the research obtain or generate genomic data?



→ If yes, answer the question below.

**a.** Will genomic data from this research be sent to a national database (for example, NIH's dbGaP database)?



→ If yes, complete the **ZIPLINE SUPPLEMENT Genomic Data Sharing** and upload it to **Zipline**.

**5.9 Whole genome sequencing.** For research involving biospecimens: Will the research include whole genome sequencing?

Whole genome sequencing is sequencing of a human germline or somatic specimen with the intent to generate the genome or exome sequence of that specimen.



#2003

- **5.10** Possible secondary use or sharing of information, specimens, or subject contact information. Is it likely that the obtained or collected information, specimens, or subject contact information will be used for any of the following:
  - Future research not described in this application (in other words, secondary research)
  - Submission to a repository, registry, or database managed by the study team, colleagues, or others for research purposes
  - Sharing with others for their own research

Please consider the broadest possible future plans and whether consent will be obtained now from the subjects for future sharing or research uses (which it may not be possible to describe in detail at this time). Answer YES even if future sharing or uses will use de-identified information or specimens. Answer NO if sharing is unlikely or if the only sharing will be through the NIH Genomic Data Sharing described in question 5.8.

Many federal grants and contracts now require data or specimen sharing as a condition of funding, and many journals require data sharing as a condition of publication. "Sharing" may include (for example): informal arrangements to share banked data/specimens with other investigators; establishing a repository that will formally share with other researchers through written agreements; or sending data/specimens to a third party repository/archive/entity such as the Social Science Open Access Repository (SSOAR), or the UCLA Ethnomusicology Archive.

| If yes, answer all of the questions below. |
|---|
| <b>a.</b> Describe what will be stored for future use, including whether any direct or indirect (e.g., subject codes) identifiers will be stored. |
| <b>b.</b> Describe what will be shared with other researchers or with a repository/database/registry, including whether direct identifiers will be shared and (for specimens) what data will be |
| released with the specimens. |
| a. Who will averse and/or manage the charing? |
| c. Who will oversee and/or manage the sharing? |
| <b>d.</b> Describe the possible future uses including limitations or restrictions (if any) on future uses or |
| d. Describe the possible future uses, including limitations or restrictions (if any) on future uses or users. As stated above, consider the broadest possible uses. |
| users. As stated above, consider the broadest possible uses. Examples: data will be used only for cardiovascular research; data will not be used for research on |

Yes  $\rightarrow$ 

#2003

| | <b>e.</b> <u>Consent</u> . Wi<br>future sharir | Il consent be obtained now from subjects for the secondary use, banking and/or |
|---|---|---|
| | No | • |
| | Yes | → If yes, be sure to include the information about this consent process in the consent form (if there is one) and in the answers to the consent questions in Section 8. |
| | | Will subjects be able to withdraw their data/specimens from secondary use, |
| | banking or sl | naring? |
| | No | → If yes, describe how, and whether there are any limitations on withdrawal. |
| | Yes | |
| | | Example: data can be withdrawn from the repository but cannot be retrieved after they are released. |
| | comply with | of for sharing or release. Confirm by checking the box that the sharing or release will UW (and, if applicable, UW Medicine) policies that require a formal agreement ipient for release of data or specimens to individuals or entities other than federal |
| | specimens (or | reements or Gatekeeping forms are used for data; Material Transfer Agreements are used for specimens plus data). Do not attach any template agreement forms; the IRB neither approves them |
| | Confir | med |
| | with already-enrolled | during the study. Describe the types of communication (if any) the research team subjects during the study. Provide a description instead of the actual materials |
| - | mail, texts, phone, or le<br>re; requests to confirm | etter reminders about appointments or about returning study materials such as a contact information. |
| througho<br>meetings | ut the course of the . SCCA subject matients come in for t | maintain communication with participating OMC provider subjects study. This will involve email communications and virtual conference tter experts would meet with subjects via bi-monthly virtual conferences heir initial visit to provide coaching on genetic counseling and testing for |
| | ntact with subjects.<br>I in the future? | Is there a plan to retain any contact information for subjects so that they can be |
| X No | | |
| Yes | be limited to the | the purpose of the future contact, and whether use of the contact information will e study team; if not, describe who else could be provided with the contact scribe the criteria for approving requests for the information. |
| | | ojects about other studies; ask subjects for additional information or medical record access part of the study proposed in this application; obtain another sample. |

# **5.13 Alternatives to participation.** Are there any alternative procedures or treatments that might be advantageous to the subjects?

If there are no alternative procedures or treatments, select "No". Examples of advantageous alternatives: earning extra class credit in some time-equivalent way other than research participation; obtaining supportive care or a standard clinical treatment from a health care provider instead of participating in research with an experimental drug.

| X | No | |
|---|-----|------------------------------------------|
| | Yes | 'es → If yes, describe the alternatives. |
| | _ | |

- **5.14 Upload to** *Zipline* all data collection forms (if any) that will be directly used by or with the subjects, and any scripts/talking points that will be used to collect the data. Do not include data collection forms that will be used to abstract data from other sources (such as medical or academic records), or video recordings.
  - **Examples**: survey, questionnaires, subject logs or diaries, focus group questions.
  - **NOTE:** Sometimes the IRB can approve the general content of surveys and other data collection instruments rather than the specific form itself. This prevents the need to submit a modification request for future minor changes that do not add new topics or increase the sensitivity of the questions. To request this general approval, use the text box below to identify the questionnaires/surveys/ etc. for which you are seeking this more general approval. Then briefly describe the scope of the topics that will be covered and the most personal and sensitive questions. The HSD staff person who screens this application will let you know whether this is sufficient or whether you will need to provide more information.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.
  - For data that will be gathered in an evolving way: This refers to data collection/questions that are not pre-determined but rather are shaped during interactions with participants in response to observations and responses made during those interactions. If this applies to the proposed research, provide a description of the process by which the data collection/questions will be established during the interactions with subjects, how the data collection/questions will be documented, the topics likely to be addressed, the most sensitive type of information likely to be gathered, and the limitations (if any) on topics that will be raised or pursued.

#### Use this text box (if desired) to provide:

- Short written descriptions of materials that cannot be uploaded, such as URLs
- A description of the process that will be used for data that will be gathered in an evolving way.
- The general content of questionnaires, surveys and similar instruments for which general approval is being sought. (See the **NOTE** bullet point in the instructions above.)

Family History Questionnaire that identifies an individual's relationship to the patient as well as their diagnosis. No PHI will be included. The purpose of this questionnaire is to identify eligible patient for genetic counseling and testing.

Patient Satisfaction Questionnaire to assess patients' experiences with genetic counseling and testing.

# **6 CHILDREN (MINORS) and PARENTAL PERMISSION**

**(6.1)Involvement of minors**. Does the research include minors (children)?

**Minor or child** means someone who has not yet attained the legal age for consent for the research procedures, as described in the applicable laws of the jurisdiction in which the research will be conducted. This may or may not be the same as the definition used by funding agencies such as the National Institutes of Health.

- In Washington State the generic age of consent is 18, meaning that anyone under the age of 18 is considered a child.
- There are some procedures for which the age of consent is much lower in Washington State.
- The generic age of consent may be different in other states, and in other countries.

| <b>X</b> No $\rightarrow$ If no, go to Section 8. | <b>No</b> $\rightarrow$ If no, go to Section 8. |
|---|---|
| Yes If yes, provide the age range of the minor subjects for this study and the legal age for consent in the study population(s). If there is more than one answer, explain. | |
| the study population(s). If there is more than one answer, explain. | |
| This means is it not possible to know the age of the subjects. For example, this may be true for some research involving social media, the Internet, or a dataset that is obtained from another researcher or from a government agency. Go to Section 8. | |
| <b>6.2 Parental permission. Parental permission</b> means actively obtaining the permission of the parents. This is <u>not</u> the same as "passive" or "opt out" permission where it is assumed that parents are allowing their children to participate because they have been provided with information about the research and have not objected or returned a form indicating they don't want their children to participate. | |
| a. Will parental permission be obtained for: | |
| All of the research procedures $\rightarrow$ Go to question 6.2b. | |
| None of the research procedures Use the table below to provide justification, and skip question 6.2b. | |
| Some of the research procedures Use the table below to identify the procedures for which parental permission will not be obtained. | |
| Be sure to consider all research procedures and plans, including screening, future contact, and sharing/banking of data and specimens for future work. | |
| Describe the procedures Children data/specimen collection (if a Group <sup>1</sup> which there will be NO pare permission <sup>2</sup> | ny) for Reason why parental Will parents be nermission will not be informed about |
| | YES NO |

Document Date & Version

Dubard-Gault 5/4/2020

11/15/2019 Version 2.2 #2003

| Table footnotes | |
|---|---|
| <ol> <li>If the answer is the same for all children groups or all procedures: collapse the answer across the groups and</li> <li>If identifiable information or biospecimens will be obtained without parent permission, any waiver granted override parents' refusal to provide broad consent (for example, through the Northwest Biotrust).</li> <li>Will parents be informed about the research beforehand even though active permission is not being obtained.</li> </ol> | by the IRB does not |
| <b>b.</b> Indicate the plan for obtaining parental permission. One or both boxes must be checked. | |
| Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably avonly one parent has legal responsibility for the care and custody of the child | vailable; or when |
| One parent, even if the other parent is alive, known, competent, reasonably available, and responsibility for the care and custody of the child. | I shares legal |
| This is all that is required for minimal risk research. | |
| If both boxes are checked, explain: | |
| <b>6.3 Children who are wards.</b> Will any of the children be wards of the State or any other agency, instit | ution or outitu? |
| No Yes → If yes, an advocate may need to be appointed for each child who is a ward. The advaddition to any other individual acting on behalf of the child as guardian or in loco same individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). The description must address the following Background and experience Willingness to act in the best interests of the child for the duration of the Independence of the research, research team, and any guardian organization. | parentis. The good points: |
| 7 ASSENT OF CHILDREN (MINORS) | |
| Go to <u>Section 8</u> if your research does not involve children (minors). | |
| 7.1 Assent of children (minors). Though children do not have the legal capacity to "consent" to particle research, they should be involved in the process if they are able to "assent" by having a study expland/or by reading a simple form about the study, and then giving their verbal choice about wheth participate. They may also provide a written assent if they are older. See WORKSHEET: Children in which a child's assent may be unnecessary or inappropriate. a. Will assent be obtained for: | plained to them<br>ther they want to |
| All research procedures and child groups $\rightarrow$ Go to guestion 7.2. | |

| | None of the resea | arch procedures and child groups | → Use the table below to provide justification, then skip to question 7.6 |
|---|---|---|---|
| Some of your research procedures and child groups | | earch procedures and child groups | Use the table below to identify the procedures for which assent will not be obtained. |
| | ure to consider all reservimens for future work. | | ng, future contact, and sharing/banking of data and |
| Ch | nildren Group¹ | Describe the procedures or data/specimen collection (if any) for which assent will NOT be obtained | Reason why assent will not be obtained |
| Table fo | | or all children groups or all procedures, collap | ose your answer across the groups and/or procedures. |
| <b>7.2 Assent process.</b> Describe how assent will be obtained, for each child group. If the research involves children of different ages, answer separately for each group. If the children are non-English speakers, include a description of how their comprehension of the information will be evaluated. | | | |
| <b>7.3 Dissent or resistance.</b> Describe how a child's objection or resistance to participation (including non-verbal indications) will be identified during the research, and what the response will be. | | | |
| <b>7.4 E-consent.</b> Will any electronic processes (email, websites, electronic signatures, etc.) be used to present assent information to subjects/and or to obtain documentation (signatures) of assent? If yes, describe how this will be done. | | | |
| | umentation of assen<br>ained? | t. Which of the following statements de | scribes whether documentation of assent will be |
| | None of the researc | ch procedures and child groups | → Use the table below to provide justification, then go to <u>question <b>7.5.b</b></u> |
| | All of the research p | procedures and child groups | → Go to question <b>7.5.a</b> , do not complete the table |
| | Some of the researc | ch procedures and/or child groups | |
| Documen | t Date & Version | | Dubard-Gault |

| _ | | Commission to be below and the control of |
|---|---|---|
| | | → Complete the table below and then to go<br>question 7.5.a |
| | Children | Describe the procedures or data/specimen collection (if any) for which assent |
| | Group <sup>1</sup> | will NOT be documented |
| <u>Table</u> | <u>footnotes</u> | |
| 1. If | the answer is the sam | e for all children groups or all procedures, collapse the answer across the groups and/or procedures. |
| ; | | ent will be documented. If the children are functionally illiterate or are not fluent in English, ion of the documentation process for them. |
| <u>C</u><br>to<br><u>C</u><br>(1 | population, and renildren who reach the hildren who were end of obtain it for the first hildren who reach the language of which the subject of the hildren who reach the subject of which the subject of the hildren who reach the subject of which the subject of the hildren who reach the subject of the subject of the subject of the subject of the subject of the hildren who reach the subject of the | standard elements of adult consent; the information should be appropriate to the age, esearch procedures. The documents should be in Word, if possible. The legal age of consent during participation in longitudinal research. The legal age of consent during participation in longitudinal research. The legal age and continue for many years: It is best practice to re-obtain assent (or set time, if it was not obtained at the beginning of their participation). The legal age of consent: Informed consent must be obtained from the now-adult subject for actions or interventions with the subjects, or (2) the continued analysis of specimens or data is identify is readily identifiable to the researcher, unless the IRB waives this requirement. The legal age of consent: The le |
| | <ul> <li>If adult cons<br/>who cannot</li> </ul> | s (if any) to obtain consent for children who reach the legal age of consent.<br>ent will be obtained from them, describe what will happen regarding now-adult subjects<br>be contacted.<br>ill not obtained or will not be possible: explain why. |
| | | uirements. (This is for information only; no answer or response is required.) Researchers are |

**7.7 Other regulatory requirements**. (This is for information only; no answer or response is required.) Researchers are responsible for determining whether their research conducted in schools, with student records, or over the Internet comply with permission, consent, and inspection requirements of the following federal regulations:

- PPRA Protection of Pupil Rights Amendment
- FERPA Family Education Rights and Privacy Act
- COPPA Children's Online Privacy Protection Act

# 8 CONSENT OF ADULTS

| 5 CONSERT OF ADOLES | |
|---|---|
| Review the following definitions | before answering the questions in this section. |
| CONSENT | is the <u>process</u> of informing potential subjects about the research and asking them whether they want to participate. It does not necessarily include the signing of a consent form. |
| CONSENT DOCUMENTATION | refers to how a subject's decision to participate in the research is documented. This is typically obtained by having the subject sign a consent form. |
| CONSENT FORM | is a document signed by subjects, by which they agree to participate in the research as described in the consent form and in the consent process. |
| ELEMENTS OF CONSENT | are specific information that is required to be provided to subjects. |
| CHARACTERISTICS OF CONSENT | <ul> <li>are the qualities of the consent process as a whole. These are: <ul> <li>Consent must be legally effective.</li> </ul> </li> <li>The process minimizes the possibility of coercion or undue influence.</li> <li>Subjects or their representatives must be given sufficient opportunity to discuss and consider participation.</li> <li>The information provided must: <ul> <li>Begin with presentation of key information (for consent materials over 2,000 words)</li> <li>Be what a reasonable person would want to have</li> <li>Be organized and presented so as to facilitate understanding</li> <li>Be provided in sufficient detail</li> <li>Not ask or appear to ask subjects to waive their rights</li> </ul> </li> </ul> |
| PARENTAL PERMISSION | is the parent's active permission for the child to participate in the research. Parental permission is subject to the same requirements as consent, including written documentation of permission and required elements. |
| SHORT FORM CONSENT | is an alternative way of obtaining written documentation of consent that is most commonly used with individuals who are illiterate or whose language is one for which translated consent forms are not available. |
| WAIVER OF CONSENT | means there is IRB approval for not obtaining consent or for not including some of the elements of consent in the consent process. NOTE: If you plan to obtain identifiable information or identifiable biospecimens without consent, any waiver granted by the IRB does not override a subject's refusal to provide broad consent (for example, the Northwest Biotrust). |
| WAIVER OF DOCUMENTATION<br>OF CONSENT | means that there is IRB approval for not obtaining written documentation of consent. |
| <b>8.1 Groups</b> Identify the groups to | which the answers in this section apply. |

X Adult subjects

Document Date & Version 11/15/2019 Version 2.2

#2003

| for all answer . "All" |
|-------------------------------|
| answer |
| . "All" |
| ens for |
| cts be with at the after ish? |
| х |
| х |

#### Table footnotes

- If the answer is the same for all groups, collapse your answer across the groups and/or procedures.
  - **b.** Describe the consent process, if consent will be obtained for any or all procedures, for any or all groups. Address groups and procedures separately if the consent processes are different.

Be sure to include:

- The location/setting where consent will be obtained
- Who will obtain consent (refer to positions, roles, or titles, not names)
- How subjects will be provided sufficient opportunity to discuss the study with the research team and consider participation

Before the start of phase 1, the SCCA study team and the potential OMC provider subjects will have a virtual meeting to discuss details of the study and prospective timeline (phase 1 and 2). Time will be allocated for the OMC providers to ask questions to ensure that there is complete understanding of the research methods, procedure, and goals. After the meeting is completed, the study's research coordinator will then email a consent information sheet to the OMC providers for review and provide a contact number if there are further questions or concerns. The OMC providers who agree to participate will send an emailed consent to the study's research coordinator.

c. Comprehension. Describe the methods that will be used to ensure or test the subjects' understanding of the information during the consent process.

The SCCA study team will host a virtual meeting with the potential OMC provider subjects to discuss the material and allow subjects to ask questions and address any concerns. After the meeting, all potential subjects will be provided a written copy of the study procedures, which will be clearly outlined and broken down by phase 1 and phase 2. The document will state the assigned responsibilities of the OMC providers and SCCA research team. The subjects will also be given a consent information sheet.

d. Influence. Does the research involve any subject groups that might find it difficult to say "no" to participation because of the setting or their relationship with someone on the study team, even if they aren't pressured to participate?

Examples: Student participants being recruited into their teacher's research; patients being recruited into their healthcare provider's research, study team members who are participants; outpatients recruited from an outpatient surgery waiting room just prior to their surgery.



No

→ If yes, describe what will be done to reduce any effect of the setting or relationship on the participation decision.

Examples: a study coordinator will obtain consent instead of the subjects' physician; the researcher will not know which subjects agreed to participate; subjects will have two days to decide after hearing about the study.

e. <u>Information provided is tailored to needs of subject population</u>. Describe the basis for concluding that the information that will be provided to subjects (via written or oral methods) is what a *reasonable member of the subject population(s)* would want to know. If the research consent materials contain a key information section, also describe the basis for concluding that the information presented in that section is that which is *most likely* to assist the selected subject population with making a decision. See <u>GUIDANCE: Key Information for Consent Materials</u>.

For example: Consultation with publications about research subjects' preferences, disease-focused nonprofit groups, patient interest groups, or other researchers/study staff with experience with the specific population. It may also involve directly consulting selected members of the study population.

The oral and written information provided to the potential OMC provider subjects covers all points that they would want to know. The information provided will explain the justification and relevance of the study, details about what participation in this study involves, and a comprehensive overview of the OMC patients' roles in the study specifically regarding medical records collection and analysis.

The key information section of the consent information sheet that SCCA will be providing includes of (1) the fact that consent is being sought for research and that participation is voluntary, (2) the purposes of the research, the expected duration of the prospective subject's participation, and the procedures to be followed in the research, (3) The most important, reasonable foreseeable risks or discomforts to the prospective subject and the benefits to the prospective subject or to others that may reasonably be expected. All of this information will assist the selected population with making a decision.

**f.** Ongoing process. For research that involves multiple or continued interaction with subjects over time, describe the opportunities (if any) that will be given to subjects to ask questions or to change their minds about participating.

The SCCA study team and participating OMC provider subjects will meet at bi-monthly virtual conferences to discuss patients. At each of these meetings, the OMC provider subjects will be given the opportunity to ask question or to change their minds about participating.

**8.3 Electronic presentation of consent information.** Will any part of the consent-related information be provided electronically for some or all of the subjects?

This refers to the use of electronic systems and processes instead of (or in addition to) a paper consent form. For example, an emailed consent form, a passive or an interactive website, graphics, audio, video podcasts. See <u>GUIDANCE: Electronic Informed Consent</u> for information about electronic consent requirements at UW.

×

**No**  $\rightarrow$  If no, skip to question 8.4

→ If yes, answer questions a through e

a. Describe the electronic consent methodology and the information that will be provided.

All informational materials must be made available to the IRB. Website content should be provided as a Word document. It is considered best practice to give subjects information about multi-page/multi-screen information that will help them assess how long it will take them to complete the process. For example, telling them that it will take about 15 minutes, or that it involves reading six screens or pages.

The consent information sheet will be sent as an electronic PDF via secure email to all OMC provider subjects.

**b.** Describe how the information can be navigated (if relevant). For example, will the subject be able to proceed forward or backward within the system, or to stop and continue at a later time?

N/A. Straightforward navigation by scrolling through the PDF document.

Document Date & Version 11/15/2019 Version 2.2 #2003 c. In a standard paper-based consent process, the subjects generally have the opportunity to go through the consent form with study staff and/or to ask study staff about any question they may have after reading the consent form. Describe what will be done, if anything, to facilitate the subject's comprehension and opportunity to ask questions when consent information is presented electronically. Include a description of any provisions to help ensure privacy and confidentiality during this process.

Examples: hyperlinks, help text, telephone calls, text messages or other type of electronic messaging, video conference, live chat with remotely located study team members.

All key points of the consent information sheet will be discussed during the initial virtual meeting with the potential OMC provider subjects and SCCA study team before the start of the study. All will be provided with the study's research coordinator's contact information in case any questions or concerns arise when reviewing the consent information sheet.

d. What will happen if there are individuals who wish to participate but who do not have access to the consent methodology being used, or who do not wish to use it? Are there alternative ways in which they can obtain the information, or will there be some assistance available? If this is a clinical trial, these individuals cannot be excluded from the research unless there is a compelling rationale.

For example, consider individuals who lack familiarity with electronic systems, have poor eyesight or impaired motor skills, or who do not have easy email or internet access.

If a participant cannot view the electronic consent form, the study's research coordinator will mail a physical copy at request. Patients who wish to participate but cannot send an emailed consent can provide verbal consent by calling the study's research coordinator (contact information is listed in the consent information sheet).

**e**. How will additional information be provided to subjects during the research, including any significant new findings (such as new risk information) If this is not an issue, explain why.

Additional information will be provided to the OMC provider subjects at the regular bi-monthly virtual conferences that will be hosted by the SCCA study team throughout the course of the study.

**8.4 Written documentation of consent.** Which of the statements below describe whether documentation of consent will be obtained? NOTE: This question does not apply to screening and recruiting procedures which have already been addressed in question 4.7.

Documentation of consent that is obtained electronically is not considered written consent unless it is obtained by a method that allows verification of the individual's signature. In other words, saying "yes" by email is rarely considered to be written documentation of consent

**a.** Is written documentation of consent being obtained for:

| X | None of the research procedures | 8.5. |
|---|---|---|
| | All of the research procedures | → Do not complete the table; go to question 8.4.b. |
| | Some of the research procedures | → Use the table below to identify the procedures for which written<br>documentation of consent will not be obtained from adult<br>subjects. |

| Adult<br>subject<br>group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which there will be NO documentation of consent | provide<br>writ<br>state<br>describ<br>rese | ney be d with a tten ment ing the arch onal)? |
|---|---|---|---|
| Phase 1 patients | Data collection of patients' medical records including clinical diagnosis and stage, pathology report features, and treatment options. OMC providers will be consenting to release the patients' medical records to the SCCA research team. | | X |
| Phase 2 patient | Data collection of patients' medical records including clinical diagnosis and stage, pathology report features, and treatment options. OMC providers will be consenting to release the patients' medical records to the SCCA research team. | | X |
| OMC<br>Providers | No documentation of consent for all aspects of this study. Per UW HSD, written documentation of consent for this minimal risk study is not needed. The SCCA study team will host a virtual meeting to offer OMC providers an opportunity to ask questions, discuss the study, and to consider participation. The SCCA study team will electronically distribute a PDF consent information sheet. | х | |
| <ul> <li>Table footnotes</li> <li>1. If the answer is the same for all adult groups or all procedures, collapse the answer across the groups and/or procedures.</li> <li>b. Electronic consent signature. For studies in which documentation of consent will be obtained: will subjects use an electronic method to provide their consent signature?</li> </ul> | | | |

- - FDA-regulated studies must use a system that complies with the FDA's "Part 11" requirements about electronic systems and records. Note that the UW-IT supported DocuSign e-signature system does not meet this requirement.
  - Having subjects check a box at the beginning of an emailed or web-based questionnaire is not considered legally

| | effectiv | re documentation of consent. |
|---|---|---|
| X | No | |
| | Yes | → If yes, describe the methodology that will be used. |
| | | See the <u>GUIDANCE: Electronic Informed Consent</u> for information about options (including the DocuSign system available through UW-IT) and requirements. |
| | | <b>b.1</b> Is this method legally valid in the jurisdiction where the research will occur? |
| | | No No |
| | | Yes $\rightarrow$ If yes, what is the source of information about legal validity? |
| | | <b>b.2</b> Will verification of the subject's identity be obtained if the signature is not personally |

witnessed by a member of the study team? Note that this is required for FDA-regulated

studies.

| No →If no, provide the rationale for why this is appropriate. Also, what would be the risks to the actual subject if somebody other than the intended signer provides the consent signature? |
|---|
| Yes → If yes, how? |
| b.3 How will the requirement be met to provide a copy of the consent information (consent<br>form) to individuals who provide an e-signature? |
| The copy can be paper or electronic and may be provided on an electronic storage device or via email. If the electronic consent information uses hyperlinks or other websites or podcasts to convey information specifically related to the research, the information in these hyperlinks should be included in the copy provided to the subjects and the website must be maintained for the duration of the entire study. |
| <b>3.5 Non-English-speaking or -reading adult subjects</b> . Will the research enroll adult subjects who do not speak English or who lack fluency or literacy in English? |
| Yes → If yes, describe the process that will be used to ensure that the oral and written information provided to them during the consent process and throughout the study will be in a language readily understandable to them and (for written materials such as consent forms or questionnaires) at an appropriate reading/comprehension level. |
| a. Interpretation. Describe how interpretation will be provided, and when. Also, describe the qualifications of the interpreter(s) – for example, background, experience, language proficiency in English and in the other language, certification, other credentials, familiarity with the research related vocabulary in English and the target language. |
| b. <u>Translations</u> . Describe how translations will be obtained for all study materials (not just consent forms). Also, describe the method for ensuring that the translations meet the UW IRB's requirement that translated documents will be linguistically accurate, at an appropriate reading level for the participant population, and culturally sensitive for the locale in which they will be used. |

ZIPLINE APPLICATION: IRB Protocol

See the <u>GUIDANCE: Electronic Informed Consent</u> for information and examples

**8.6 Barriers to written documentation of consent.** There are many possible barriers to obtaining written documentation of consent. Consider, for example, individuals who are functionally illiterate; do not read English well; or have sensory or motor impairments that may impede the ability to read and sign a consent form. a. Describe the plans (if any) for obtaining written documentation of consent from potential subjects who may have difficulty with the standard documentation process (that is, reading and signing a consent form). Skip this question if written documentation of consent is not being obtained for any part of the research. Examples of solutions: Translated consent forms; use of the Short Form consent process; reading the form to the person before they sign it; excluding individuals who cannot read and understand the consent form. N/A. Written documentation of consent is not being obtained for any part of the research. 8.7) Deception. Will information be deliberately withheld, or will false information be provided, to any of the subjects? Note: "Blinding" subjects to their study group/condition/arm is not considered to be deception, but not telling them ahead of time that they will be subject to an intervention or about the purpose of the procedure(s) is deception. No → If yes, describe what information and why. Yes Example: It may be necessary to deceive subjects about the purpose of the study (describe why). a. Will subjects be informed beforehand that they will be unaware of or misled regarding the nature or purposes of the research? (Note: this is not necessarily required.) No Yes **b.** Will subjects be debriefed later? (Note: this is not necessarily required.) No → If yes, describe how and when this will occur. Upload any debriefing materials, Yes including talking points or a script, to **Zipline**. (8.8) Cognitively impaired adults, and other adults unable to consent. Will such individuals be included in the research? Examples: individuals with Traumatic Brain Injury (TBI) or dementia; individuals who are unconscious, or who are significantly intoxicated. No  $\rightarrow$  If no, go to question 8.9. Yes → If yes, answer the following questions. **a.** Rationale. Provide the rationale for including this population.

| b. Capacity for consent / decision making capacity. Describe the process that will be used to<br>determine whether a cognitively impaired individual is capable of consent decision making<br>with respect to the research protocol and setting. |
|---|
| b.1. If there will be repeated interactions with the impaired subjects over a time period when cognitive capacity could increase or diminish, also describe how (if at all) decision-making capacity will be re-assessed and (if appropriate) consent obtained during that time. |
| c. <u>Permission</u> (surrogate consent). If the research will include adults who cannot consent for<br>themselves, describe the process for obtaining permission ("surrogate consent") from a legally<br>authorized representative (LAR). |
| For research conducted in Washington State, see the <b>GUIDANCE: Legally Authorized Representative</b> to learn which individuals meet the state definition of "legally authorized representative". |
| d. <u>Assent</u> . Describe whether assent will be required of all, some, or none of the subjects. If some, indicate which subjects will be required to assent and which will not (and why not). Describe any process that will be used to obtain and document assent from the subjects. |
| <ul> <li>e. <u>Dissent or resistance</u>. Describe how a subject's objection or resistance to participation<br/>(including non-verbal) during the research will be identified, and what will occur in response.</li> </ul> |
| <b>8.9 Research use of human fetal tissue obtained from elective abortion.</b> Federal and UW Policy specify some requirements for the consent process. If you are conducting this type of research, check the boxes to confirm these requirements will be followed. Informed consent for the donation of fetal tissue for research use will be obtained by someone other than |
| the person who obtained the informed consent for abortion. |
| Informed consent for the donation of fetal tissue for research use will be obtained after the informed consent for abortion. |
| Participation in the research will not affect the method of abortion. |
| No enticements, benefits, or financial incentives will be used at any level of the process to incentivize abortion or the donation of human fetal tissue. |
| The informed consent form for the donation of fetal tissue for use in research will be signed by both the |

woman and the person who obtains the informed consent.

- **8.10 Consent-related materials**. Upload to *Zipline* all consent scripts/talking points, consent forms, debriefing statements, Information Statements, Short Form consent forms, parental permission forms, and any other consent-related materials that will be used. Materials that will be used by a specific site should be uploaded to that site's **Local Site Documents** page.
  - <u>Translations must be submitted and approved before they can be used</u>. However, we strongly encourage you to wait to provide them until the IRB has approved the English versions.
  - <u>Combination forms</u>: It may be appropriate to combine parental permission with consent, if parents are subjects as well as providing permission for the participation of their children. Similarly, a consent form may be appropriately considered an assent form for older children.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. URLs (website addresses) may also be provided, or written descriptions of websites. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.

### 9 PRIVACY AND CONFIDENTIALITY

**9.1 Privacy protections.** Describe the steps that will be taken, if any, to address possible privacy concerns of subjects and potential subjects.

Privacy refers to the sense of being in control of access that others have to ourselves. This can be an issue with respect to recruiting, consenting, sensitivity of the data being collected, and the method of data collection. Examples:

- Many subjects will feel a violation of privacy if they receive a letter asking them to participate in a study because they
  have \_\_\_\_ medical condition, when their name, contact information, and medical condition were drawn from medical
  records without their consent. Example: the IRB expects that "cold call" recruitment letters will inform the subject
  about how their information was obtained.
- Recruiting subjects immediately prior to a sensitive or invasive procedure (e.g., in an outpatient surgery waiting room) will feel like an invasion of privacy to some individuals.
- Asking subjects about sensitive topics (e.g. details about sexual behavior) may feel like an invasion of privacy to some individuals.

This is a quality improvement research study that intends to improve the standard processes of care for OMC cancer patients regarding genetic counseling and genetic testing. All collection and review of patients' information and medical records will be part of their clinical care and screening. The patients' information will not be used for any type of enrollment or recruitment. The OMC providers (study's subjects) will grant permissions for the release of their patients' medical records to the SCCA study team by reviewing a consent information sheet and sending emailed consent to the study's research coordinator.

| subjects be used in pul | duals in publications and presentations. Will potentially identifiable information about olications and presentations, or is it possible that individual identities could be inferred from published or presented? |
|---|---|
| X No<br>Yes → If yes, wi | Il subject consent be obtained for this use? |
| No | → If no, describe the steps that will be taken to protect subjects (or small groups of subjects) from being identifiable. |
| Document Date & Version | Dubard-Gault |

9.3 State mandatory reporting. Each state has reporting laws that require some types of individuals to report some kinds of abuse, and medical conditions that are under public health surveillance. These include:

Child abuse
Abuse, abandonment, neglect, or financial exploitation of a vulnerable adult
Sexual assault
Serious physical assault
Medical conditions subject to mandatory reporting (notification) for public health surveillance

Are you or a member of the research team likely to learn of any of the above events or circumstances while

Are you or a member of the research team likely to learn of any of the above events or circumstances while conducting the research **AND** feel obligated to report it to state authorities?

| X | No |
|---|-----|
| | Yes |

→ If yes, the UW IRB expects subjects to be informed of this possibility in the consent form or during the consent process, unless you provide a rationale for not doing so:

**9.4 Retention of identifiers and data.** Check the box below to indicate assurance that any identifiers (or links between identifiers and data/specimens) and data that are part of the research records will not be destroyed until after the end of the applicable records retention requirements (e.g. Washington State; funding agency or sponsor; Food and Drug Administration). If it is important to say something about destruction of identifiers (or links to identifiers) in the consent form, state something like "the link between your identifier and the research data will be destroyed after the records retention period required by state and/or federal law."

This question can be left blank for conversion applications (existing paper applications that are being "converted" into a Zipline application.)

See the "Research Data" sections of the following website for UW Records management for the Washington State research rectords retention schedules that apply in general to the UW (not involving UW Medicine data): <a href="http://f2.washington.edu/fm/recmgt/gs/research?title=R">http://f2.washington.edu/fm/recmgt/gs/research?title=R</a>

See the "Research Records and Data" information in Section 8 of this document for the retention schedules for UW Medicine Records: https://www.uwmedicine.org/recordsmanagementuwm-records-retention-schedule.pdf



**9.5 Certificates of Confidentiality**. Will a federal Certificate of Confidentiality be obtained for the research data? *NOTE: Answer "No" if the study is funded by NIH or the CDC, because all NIH-funded and CDC-funded studies automatically have a Certificate.* 



- 9.6 Data and specimen security protections. Identify the data classifications and the security protections that will be provided for all sites where data will be collected, transmitted, or stored, referring to the ZIPLINE GUIDANCE:

  Data and Security Protections for the minimum requirements for each data classification level. It is not possible to answer this question without reading this document. Data security protections should not conflict with records retention requirements.
  - **a.** Which level of protections will be applied to the data and specimens? If more than one level will be used, describe which level will apply to which data and which specimens and at which sites.

Level 4

- b. Use this space to provide additional information, details, or to describe protections that do not fit into one of the levels. If there are any protections within the level listed in 9.6.a which will not be followed, list those here, including identifying the sites where this exception will apply.
  - All level 4 data collected by OMC will be part of their standard processes of care. The only individual outside of OMC to have access to the identified data will be the study's research coordinator at SCCA. The research coordinator will follow all user, device, server, and data transmission guidelines. Any information provided to the SCCA subject matter experts will be deidentified.

# **10 RISK / BENEFIT ASSESSMENT**

- (10.1)Anticipated risks. Describe the <u>reasonably foreseeable</u> risks of harm, discomforts, and hazards to the subjects and others of the research procedures. For each harm, discomfort, or hazard:
  - Describe the magnitude, probability, duration, and/or reversibility of the harm, discomfort, or hazard, AND
  - Describe how the risks will be reduced or managed. Do not describe data security protections here, these are already described in Question 9.6.
  - Consider possible physical, psychological, social, legal, and economic harms, including possible negative effects on financial standing, employability, insurability, educational advancement or reputation. For example, a breach of confidentiality might have these effects.
  - Examples of "others": embryo, fetus, or nursing child; family members; a specific group.
  - Do not include the risks of non-research procedures that are already being performed.
  - If the study design specifies that subjects will be assigned to a specific condition or intervention, then the condition or intervention is a research procedure - even if it is a standard of care.
  - Examples of mitigation strategies: inclusion/exclusion criteria; applying appropriate data security measures to prevent unauthorized access to individually identifiable data; coding data; taking blood samples to monitor something that indicates drug toxicity.
  - As with all questions on this application, you may refer to uploaded documents.

Participation in this study involves a time commitment from the OMC provider subjects in which they are required to designate time from their schedule to participate in bi-monthly virtual conferences. If a participant decides to implement the coaching from SCCA in their clinical care, time will be required to discuss genetic counseling and testing with their eligible patients, ordering genetic testing, and allocating extra time at patient follow-up visits to review genetic results. This time commitment may cause stress in the OMC provider subjects because it will likely require them to change how they manage their schedules.

This study requires OMC provider subjects to grant permissions to SCCA to collect their patients' medical records, which may pose security concerns and a breach of confidentiality for their patients.

(10.2) Reproductive risks. Are there any risks of the study procedures to men and women (who are subjects, or partner of subjects) related to pregnancy, fertility, lactation or effects on a fetus or neonate?

Examples: direct teratogenic effects; possible germline effects; effects on fertility; effects on a woman's ability to continue a pregnancy; effects on future pregnancies.

| X | No |
|---|-----|
| | Yes |

→ If no go to question 10.3

→ If yes, answer the following questions:

a. Risks. Describe the magnitude, probability, duration and/or reversibility of the risks.

Version 2.2

| | Examples: inform the subjects about the risks and how to minimize them; require a and during the study; require subjects to use contraception; advise subjects about b ova. | |
|---|---|---|
| | If the use of contraception will be required: describe the allowable methods and the contraception must be used. | time period when |
| | c. Pregnancy. Describe what will be done if a subject (or a subject's partne | r) becomes pregnant |
| | For example; will subjects be required to immediately notify study staff, so that the discontinue or modified, or for a discussion of risks, and/or referrals or counseling? | study procedures can be |
| reaction calle<br>received gad<br>allergic react<br>a. Describe h | nagement. Answer this question only if the subjects will receive MRI scans. A railed nephrogenic systemic fibrosis (NSF) has been observed in individuals with kid olinium-based contrast agents (GBCAs) for the scans. Also, a few healthy individuals tion to GBCAs. Inow the renal function of subjects will be assessed prior to MRI scans and how to exclude subjects at risk for NSF. | dney disease who<br>duals have a severe |
| N/A, sub | ojects will not receive MRI scans | |
| | he protocol for handling a severe allergic reaction to the GBCA or any other me<br>tergency during the MRI scan, including who will be responsible for which action | |
| N/A, sub | jects will not receive MRI scans | |
| 10.4 Unforeseeal | ble risks. Are there any research procedures that may have risks that are curren | tly unforeseeable? |
| Example: usin | g a drug that hasn't been used before in this subject population. | |
| X No | | |
| Yes | → If yes, identify the procedures. | |
| patients are | o will be under regional or general anesthesiology. Will any research procedur under general or regional anesthesia, or during the 3 hours preceding general or non-research reasons)? | |
| Yes | → If yes, check all the boxes that apply. | |
| | Administration of any drug for research purposes | |
| | Inserting an intra-venous (central or peripheral) or intra-arterial line fo | r research purposes |
| | Obtaining samples of blood, urine, bone marrow or cerebrospinal fluid purposes | for research |
| Document Date & Ve | rsion | Dubard-Gault |
| 11/15/2019 | ZIPLINE APPLICATION: IRB Protocol | 5/4/2020<br>Version 1 |

**b. Steps to minimize risk**. Describe the specific steps that will be taken to minimize the

magnitude, probability, or duration of these risks.

| Obtaining a research sample from tissue or organs that would not otherwise be removed during surgery |
|---|
| Administration of a radio-isotope for research purposes** |
| Implantation of an experimental device |
| Other manipulations or procedures performed solely for research purposes (e.g., experimental liver dialysis, experimental brain stimulation) |
| If any of the boxes are checked: Provide the name and institutional affiliation of a physician anesthesiologist who is a member of the research team or who will serve as a safety consultant about the interactions between the research procedures and the general or regional anesthesia of the subject-patients. If the procedures will be performed at a UW Medicine facility or affiliate, the anesthesiologist must be a UW faculty member, and the Vice Chair of Clinical Research in the UW Department of Anesthesiology and Pain Medicine must be consulted in advance for feasibility, safety and billing. |

10.6 Data and Safety Monitoring. A Data and Safety Monitoring Plan (DSMP) is required for clinical trials (as defined by NIH). If required for this research, or if there is a DSMP for the research regardless of whether it is required, upload the DSMP to *Zipline*. If it is embedded in another document being uploading (for example, a Study Protocol) use the text box below to name the document that has the DSMP. Alternatively, provide a description of the DSMP in the text box below.

The OMC provider subjects will be given detailed instructions (both written and verbal) on how to collect relevant patient data and send electronically to the study's research coordinator (via secure email). Once received by the study's research coordinator, the data will be stored in a secured J-Drive folder within the SCCA network. The research coordinator will randomly assign all identified patient data to a unique participant ID before distributing to SCCA subject matter experts (cancer geneticist and/or genetic counselor) for review. For the bi-monthly conference meetings in which the SCCA subject matter experts review patients' medical records, the study's research coordinator will order the patients for discussion (OMC providers will receive the meeting agendas that lists the patient discussion order which will include patient PHI. SCCA subject matter experts will also receive meeting agendas that lists the same patient discussion order but will only have access to the unique participant ID and no PHI).

**10.7 Un-blinding.** If this is a double-blinded or single-blinded study in which the participant and/or relevant study team members do not know the group to which the participant is assigned: describe the circumstances under which un-blinding would be necessary, and to whom the un-blinded information would be provided.

N/A. This is not a double-blinded or single-blinded study.

<sup>\*\*</sup> If the box about radio-isotopes is checked: the study team is responsible for informing in advance all appropriate clinical personnel (e.g., nurses, technicians, anesthesiologists, surgeons) about the administration and use of the radio-isotope, to ensure that any personal safety issues (e.g., pregnancy) can be appropriately addressed. This is a condition of IRB approval.

| <b>10.8 Withdrawal of participants.</b> If applicable, describe the anticipated circumstances under which participants will be withdrawn from the research without their consent. Also, describe any procedures for orderly withdrawal of a |
|---|
| participant, regardless of the reason, including whether it will involve partial withdrawal from procedures and any intervention but continued data collection or long-term follow-up. |
| (10.9) Anticipated direct benefits to participants. If there are any direct research-related benefits that some or all individual participants are likely to experience from taking part in the research, describe them below: |
| Do not include benefits to society or others, and do not include subject payment (if any). Examples: medical benefits such as laboratory tests (if subjects receive the results); psychological resources made available to participants; training or education that is provided. |
| This research will improve patient access to genetic testing which would enable us to identify if there are any previously undetected genetic predispositions in a patient's family. As a result, we can offer participation in cancer screening, surveillance, and prevention programs for family members at risk of cancer to decrease their risk to as close to zero as possible. Overall, this study will improve utilization of genetic counseling and testing amongst OMC providers caring for their cancer patients. |
| 10.10 Return of individual research results. |
| In this section, provide your plans for the return of individual results. An "individual research result" is any information collected, generated or discovered in the course of a research study that is linked to the identity of a research participant. These may be results from screening procedures, results that are actively sought for purposes of the study, results that are discovered unintentionally, or after analysis of the collected data and/or results has been completed. |
| See the <u>GUIDANCE Return of Individual Results</u> for information about results that should and should not be returned, validit of results, the Clinical Laboratory Improvement Amendment (CLIA), consent requirements and communicating results. |
| a. Is it anticipated that the research will produce any individual research results that are clinically actionable |
| "Clinically actionable" means that there are established therapeutic or preventive interventions or other available actions that have the potential to change the clinical course of the disease/condition, or lead to an improved health outcome. |
| In general, every effort should be made to offer results that are clinically actionable, valid and pose life-threatening severe health consequences if not treated or addressed quickly. Other clinically actionable results should be offered in this can be accomplished without compromising the research. X No |
| Yes → If yes, answer the following questions (a.1-a.3). |
| a.1. Describe the clinically actionable results that are anticipated and explain which results<br>if any, could be urgent (i.e. because they pose life-threatening or severe health<br>consequences if not treated or addressed quickly). |
| Examples of urgent results include very high calcium levels, highly elevated liver function test result positive results for reportable STDs. |
| a.2. Explain which of these results will be offered to subjects. |
| Document Date & Version Dubard-Gat |

| • | plain which results will <u>not</u> be offered to subjects and provide the rationale for not |
|---|---|
| offer | ring these results. |
| Reason | s not to offer the results might include: |
| • | There are serious questions regarding validity or reliability |
| • | Returning the results has the potential to cause bias |
| • | There are insufficient resources to communicate the results effectively and appropriately |
| • | Knowledge of the result could cause psychosocial harm to subjects |

| b. | . What is the plan (i | if anv) for | offering subject | ts any results tha | at are not clinically | actionable? |
|---|---|---|---|---|---|---|

Examples: non-actionable genetic results, clinical tests in the normal range, experimental and/or uncertain results.

| X | No | |
|---|---|---|
| | Yes | → If yes, explain which results will be offered to subjects and provide the rationale for offering these results. |

c. Describe the validity and reliability of any results that will be offered to subjects.

The IRB will consider evidence of validity such as studies demonstrating diagnostic, prognostic, or predictive value, use of confirmatory testing, and quality management systems.

The results that will be offered to the OMC provider subjects will be reliable due to the consistent, uniform processes in data collection and recommendation that will be followed throughout the entire course of this study. The results will be valid because the reporting of the numbers of patients meeting criteria, referrals for genetic counseling/testing, completed genetics appointments, and genetic testing results, will be recorded and tracked by the same research coordinator.

**d**. Describe the process for communicating results to subjects and facilitating understanding of the results. In the description, include who will approach the participant with regard to the offer of results, who will communicate the result (if different), the circumstances, timing, and communication methods that will be used.

Results will be communicated to the OMC provider subjects at the end of phase 1 and phase 2. The SCCA study team and subjects will meet to discuss the number of patients seen who were eligible for genetic testing, number of those patients who were referred for genetic counseling/testing, the number of those patients who complete a genetics appointment, and the number of those patients who chose to undergo genetic testing. The OMC provider subjects will also be sent this data for their review in order to assess their current clinic processes.

**e**. Describe any plans to share results with family members (e.g. in the event a subject becomes incapacitated or deceased).

N/A

**f**. Check the box to indicate that any plans for return of individual research results have been described in the consent document. If there are no plans to provide results to participants, this should be stated in the consent form.

See the **GUIDANCE Return of Individual Results** for information about consent requirements.

| <br>1 |
|-----------|
| Confirmed |

**10.11 Commercial products or patents**. Is it possible that a commercial product or patent could result from this study?

| X No | 0 |
|------|---|
|------|---|

#2003

Document Date & Version

11/15/2019

Version 2.2

ZIPLINE APPLICATION: IRB Protocol

| | Yes → If yes, describe whether subjects might receive any remuneration/compensation and, if yes, how the amount will be determined. |
|---|---|
| 11 E | ECONOMIC BURDEN TO PARTICIPANTS |
| | <b>Financial responsibility for research-related injuries.</b> Answer this question only if the lead researcher is <u>not</u> a UW student, staff member, or faculty member whose primary paid appointment is at the UW. |
| | For each institution involved in conducting the research: Describe who will be financially responsible for research-related injuries experienced by subjects, and any limitations. Describe the process (if any) by which participants may obtain treatment/compensation. |
| | N/A. The lead research is a UW staff member whose primary paid appointment is at the UW. |
| | <b>Costs to subjects</b> . Describe any research-related costs for which subjects and/or their health insurance may be responsible (examples might include: CT scan required for research eligibility screening; co-pays; surgical costs when a subject is randomized to a specific procedure; cost of a device; travel and parking expenses that will not be reimbursed). |
| 11.3 | Reimbursement for costs. Describe any costs to subjects that will be reimbursed (such as travel expenses). |

### **12 RESOURCES**

- **12.1) Faculty Advisor.** (For researchers who are students, fellows, or post-docs.) Provide the following information about the faculty advisor.
  - Advisor's name
  - Your relationship with your advisor (for example: graduate advisor; course instructor)
  - Your plans for communication/consultation with your advisor about progress, problems, and changes.

N/A

**12.2 UW Principal Investigator Qualifications**. Upload a current or recent Curriculum Vitae (CV), Biosketch (as provided to federal funding agencies), or similar document to the Local Site Documents page in Zipline. The purpose of this is to address the PI's qualifications to conduct the proposed research (education, experience, training, certifications, etc.).

For help with creating a CV, see <a href="http://adai.uw.edu/grants/nsf">http://adai.uw.edu/grants/nsf</a> biosketch template.pdf</a> and <a href="https://education.uwmedicine.org/student-affairs/career-advising/year-4/residency-applications/curriculum-vitae/">https://education.uwmedicine.org/student-affairs/career-advising/year-4/residency-applications/curriculum-vitae/</a>

X The CV will be uploaded.

#2003

**12.3 UW Study team qualifications**. Describe the qualifications and/or training for each <u>UW</u> study team member to fulfill their role on the study and perform study procedures. (You may be asked about non-UW study team members during the review; they should not be described here.) You may list these individuals by name, however if you list an individual by name, you will need to modify this application if that individual is replaced.

Page 44 of 46

Document Date & VersionDubard-Gault11/15/20195/4/2020Version 2.2ZIPLINE APPLICATION: IRB ProtocolVersion 1

Alternatively, you can describe study <u>roles</u> and the qualifications and training the PI or study leadership will require for any individual who might fill that role. The IRB will use this information to assess whether risks to subjects are minimized because study activities are being conducted by properly qualified and trained individuals.

Describe: The role (or name of person), the study activities they will perform, and the qualifications or training that are relevant to performing those study activities.

### **Examples:**

<u>Research Study Coordinator:</u> Obtain consent, administer surveys, blood draw. Will have previous experience coordinating clinical research and be a certified phlebotomist in WA.

<u>Undergraduate Research Assistant:</u> Obtain consent, perform all study procedures. Will have had coursework in research methods, complete an orientation to human subjects protections given by the department, and will receive training from the PI or the graduate student project lead on obtaining consent and debriefing subjects. <u>Acupuncturist:</u> Perform acupuncture procedures and administer surveys. Must be licensed with WA State DoH and complete training in administering research surveys given by the project director, an experienced survey researcher.

<u>Co-Investigator:</u> Supervise MRI and CT scan procedures and data interpretation, obtain consent. MD, specialty in interventional radiology and body imaging. 5-years clinical research experience.

Research Study Coordinator (Lauren Santos): Will obtain and securely store all study data and distribute appropriately to SCCA subject matter experts for review, facilitate communications between OMC and SCCA, participate in data analysis of study's result. Has completed the Human Subjects Learners and Good Clinical Practice and ICH (GCP) certification from the Collaborative Institutional Training Initiative (CITI). Has prior experience with data analysis and data visualization through UW's Healthcare Analytics certificate program. Completed Microsoft Excel workshops and data organization/data science classes through Fred Hutch Learning.

| adequately trained and informed about the research procedures and requirements (including any changes) as well as their research-related duties and functions. |
|---|
| There is no study team. |
| The study team will meet bi-monthly to discuss and debrief research procedures and requirements as well as their research-related duties and function. The study team will also regularly meet with OMC to ensure complete understanding of data collection and distribution processes. |
| 13 OTHER APPROVALS, PERMISSIONS, and REGULATORY ISSUES |

13.1) Approvals and permissions. Identify any other approvals or permissions that will be obtained. For example: from

a school, external site/organization, funding agency, employee union, UW Medicine clinical unit.

Do not attach the approvals and permissions unless requested by the IRB.

N/A

| | Financial Conflict of Interest. Does any UW member of the team have ownership or other Significant Fin Interest (SFI) with this research as defined by <a href="https://example.com/linearing/linearing-new-maps-scripts">UW policy GIM 10</a> ? | |
|---|---|---|
| X No<br>Yes | → If yes, has th proposed res | e Office of Research made a determination regarding this SFI as it pertains to the search? |
| No | | → If no, contact the Office of Research (206.616.0804, <a href="mailto:research@uw.edu">research@uw.edu</a> ) for guidance on how to obtain the determination |
| | Yes | → If yes, upload the Conflict Management Plan for every UW team member who has a FCOI with respect to the research, to <i>Zipline</i> . If it is not yet available, use the text box to describe whether the Significant Financial Interest has been disclosed already to the UW Office of Research and include the FIDS Disclosure ID if available. |